CLINICAL TRIAL: NCT04444271
Title: Prospective, Randomized Phase 2 Clinical Trial of Mesenchymal Stem Cells(MSCs) for the Treatment of Coronavirus Disease 2019(COVID-19)
Brief Title: Mesenchymal Stem Cell Infusion for COVID-19 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Zaineb Akram (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Zaineb Akram, Research officer, National Institute of Blood and Marrow Transplant (NIBMT), Pakistan
Organization: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBMT-MSc-COVID-2020
Record Dates: First submitted 2020-05-27; First posted 2020-06-23 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: Coronavirus; Mesenchymal Stem Cells; Survival
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells (Experimental): 10 patients will be given mesenchymal stem cells at dose 2x10^6 cells/kg MSCs on days 1 and day 7 (if needed) in addition to standard care
  Interventions: Drug: Mesenchymal stem cells
- Placebo (Placebo Comparator): Only supportive care will be given to 10 patients
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesenchymal stem cells — 1. Frozen MSCs will be resuspended in 100ml normal saline for immediate use and given intravenously. The patients should be pre-medicated to avoid allergic reactions to third party MSCs. Each patient in Experimental arm will be given 2 x 106 cells/kg will be administered on day 1,7 in addition to supportive care
  Other Names: MSCs
  Arms: Mesenchymal stem cells
Other: Placebo — 100 ml of normal saline will be given intravenously to control arm
  Arms: Placebo

SUMMARY:
Since the outbreak of coronavirusdisease2019(COVID-19), many researchers in China have carried out/published clinical trials on treatment based on Western medicine, traditional Chinese medicine or a combination of the two. Trials on treatment modalities have mainly used antivirals, interferon, glucocorticoids in addition to traditional Chinese medicine. There are also clinical trials exploring hydroxyquinoline/chloroquine sulphate, immunoglobulins, Vitamin-C, washed microbiota, nebulized interferon, teicoplanin as well as Mesenchymal stem cells. However, most of these trials were small (median sample size 100) and the bulk of potential therapeutic strategies remain in the experimental phase and currently there is no eﬀective speciﬁc antiviral with high-level evidence.The aim of this study is assess the efficacy of MSCs as an add-on therapy to standard supportive treatment for patients with moderate/severe COVID-19.

DETAILED DESCRIPTION:
All patients will receive 2x10^6 cells/kg on days 1 and day 7 (if needed). The study will be divided in 2 phases. In the first phase, 10 patients will be included and randomized to 2 groups (5 Treatment arm; 5 Control Arm) and receive 2 x10^6 cells/kg MSCs on days 1 and 7 in addition to standard care. Thereafter, the trial committee will meet and evaluate all collected safety and efficacy information to decide about crossover of Control arm to treatment arm if patient deteriorates clinically while in Control arm. Then, 10 new subjects will be included in the study and treated according to protocol.

Preparation of MSCs doses MSCs will be isolated from bone marrow harvested cells. About 50ml bone marrow will be collected from iliac crest using aseptic technique in syringes primed with anticoagulant. The collected sample will be diluted with Phosphate Buffer Saline (PBS) and MSCs will be separated using density gradient centrifugation. After resuspension the cells will be seeded at a fixed concentration of 100,000 cells/cm2 in specially designed flasks and incubated at 37oC in 5% carbondioxide (CO2). Medium will be changed after every third day till harvesting of MSCs from the flasks. Once confluent (approximately day 20) the cells will be harvested with sterile techniques using Trypsin- Ethylenediaminetetraacetic acid ( EDTA ) solution. The prepared cells can either be stored in 50ml cryogenic vials for future use or infused immediately.

Patient Selection and MSCs demand Patient for MSCs and Control arm will be selected by multidisciplinary team (MDT) comprising Critical Care Specialist, Pulmonologist, Infectious Disease Specialist, Clinical Hematologist.

1. Demand for MSCs will be initiated on pre-designated forms , signed by Critical care Specialist Clearly indicating indication of MSCs.
2. Request form will be sent Stem Cell Lab.
3. Incharge stem Cell Lab will authorize issuance of the MSCs dose.
4. Stem Cell Lab will issue the dose Administration of MSCs

1. Experimental arm: Frozen MSCs will be resuspended in 100ml normal saline for immediate use and given intravenously. The patients should be pre-medicated to avoid allergic reactions to third party MSCs. Each patient in Experimental arm will be given 2 x 106 cells/kg will be administered on day 1,7 in addition to supportive care 2. Control Arm: Will be Continued on supportive care

Proposed usage:

Because of the very limited availability of MSCs, their usage has to be rationalized by MDT comprising of pulmonologist, critical care specialist and clinical haematologist and Infectious disease specialist.There is not enough evidence to put forth therapeutic recommendations however, treatment decisions can be made on case to case basis after MDT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 10years
2. Laboratory confirmation of COVID19 infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source; and
3. Moderate illness: In compliance with the 2019-coronavirus pneumonia diagnosis standard [according to the novel coronavirus infection pneumonia diagnosis and treatment program (Trial Implementation Version 6) issued by the National Health and Medical Commission, and world health organization (WHO) 2019 new coronavirus guidelines standards]: (A) increased breathing rate (≥30 beats / min), difficulty breathing, cyanosis of the lips; (B) in resting state, means oxygen saturation ≤93%; (C) partial pressure of arterial oxygen (PaO2) / Fraction of inspired oxygen (FiO2) ≤300 mmHg (1mmHg = 0.133kPa);
4. Critically ill : Respiratory failure, Septic Shock, muti-organ dysfunction syndrome (MODS)

Exclusion Criteria:

1. Patients with systemic autoimmune diseases
2. Not consenting for clinical trial
3. Those declared not for resuscitation due to underlying comorbid or current critical condition

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 30 days post intervention
  Assessment of Overall survival at 30 days post intervention

SECONDARY OUTCOMES:
Clinical improvement | 30 days
  days required for oxygen support independence after intervention
Time of COVID19 PCR negativity | day 1,3,7,10, 14
  PCR testing to check PCR negativity
Radiological improvement (day 15 and day 30 assessment) | day 15 and day30
  Computed tomography Chest assesment will be done to assess improvment in radiological findings of COVID-19
days required to discharge from hospital | 30 days post admission
  number of days required for discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: xanab akram, Study Chair — NIBMT
Locations (1):
- NIBMT, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No